CLINICAL TRIAL: NCT06584604
Title: Calibration of Esophageal Balloon Catheter in Spontaneous and Mandatory Mechanical Ventilation (PESCA)
Brief Title: Calibration of Esophageal Balloon Catheter in Spontaneous and Mandatory Mechanical Ventilation
Acronym: PESCA
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Abraham Schoe, MD, PhD., MD, PhD, Principal Investigator, Leiden University Medical Center
Other Study IDs: NL83335.058.24
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Unit; Mechanical Ventilation; Critical Illness
Keywords: Esophageal Pressure; Esophageal Balloon Catheter; Transpulmonary Pressure; Mandatory Ventilation; Support Ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
Calibration of the esophageal balloon catheter (Pes catheter) is important for the right measurement of the esophageal pressure (Pes) and subsequent interpretation of the derived transpulmonary pressures during mechanical ventilation. Both relative changes and absolute values of Pes can be affected by inappropriate filling of the esophageal balloon and by the elastance of the esophagus wall. Therefore one should calibrate the balloon to determine the best filling pressure. Calibration of the Pes catheter has only been validated in mandatory ventilation but not in support modes in which the patient triggers the ventilator and is supported by the mechanical ventilator. Because the forces in the thoracic cage behave differently in comparison with a controlled mode, it is to be expected that the calibration process in a support mode yields different filling volumes in comparison with the calibration process in a controlled mode. This would lead to a more reliable filling volume in support mechanical ventilation and a more reliable derivation of transpulmonary pressure and therefore to a better treatment of patients.

DETAILED DESCRIPTION:
In mechanical ventilation the esophageal pressure (Pes) is used to calculate the transpulmonary pressure (PL). The transpulmonary pressure is used to set the positive end expiratory pressure (PEEP) and the inspiratory pressure. In spontaneous mechanical ventilation the transpulmonary pressure swing (which is the difference between the maximum and minimum transpulmonary pressure) is used as a measure of patient effort. Too much patient effort is perhaps detrimental in patients with early, severe ARDS, leading to additional lung damage and possibly a prolonged ICU stay.

The Pes is measured using a separate or integrated (feeding tube and Pes catheter) esophageal balloon catheter. The catheter is placed in the right position and has to be inflated to produce a readable pressure signal. The Pes balloon needs calibration before measurement to be sure that the readings are trustworthy. When calibrating one should take the compliance of the esophagus into account, together with the calibration curve, and with that, the filling volume of the patient changes from patient to patient. A calibration study of the Pes catheter has only been performed in passive mechanically ventilated patients, i.e. in patients without any breathing efforts.

In spontaneous breathing patients who still needs support from the ventilator, the forces within the thorax differ considerably in comparison with passive patients. When initiating a breath the diaphragm of the patient will move downwards and the Pes will become negative. In passive patient the ventilator initiates the breath and the diaphragm will be pushed downwards but the Pes will become more positive. It is probable that the calibration methods used in passive patients is not feasible in patients who exhibit a breathing effort. It is therefore necessary to study the calibration of the esophageal balloon catheter in patients that breath spontaneously with the support of a mechanical ventilator.

The hypothesis is that the calibration method, and therefore the filling pressure of the balloon is different from the values when the patient would be ventilated in a passive mode. Wrong calibration leads to wrong values, which could possibly lead to wrong interpretation of the obtained values with possible harm for the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Mechanically ventilated in spontaneous mode.
* Sedated (Richmond Agitation Sedation Scale (RASS) between -3 and -5).
* Pes catheter in situ according to the protocol used in the LUMC (Insertion of a Pes catheter is mandatory if it is suspected that te patient will be ventilated for more than 24 hrs.).

Exclusion Criteria:

* Medical condition that excludes the placement of a Pes catheter.
* Allergic reaction against rocuronium in the past.
* Pregnant.
* RASS > -3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients who are on mechanical ventilation with a esophageal balloon catheter in situ according to the current LUMC protocol. Expected mechanical ventilation time > 24 hrs. RASS between -3 and -5;
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressures (in cmH2O) measured by the balloon catheter at different filling volumes (in ml) | 45 minutes
  To obtain a calibration method for the oesophageal balloon catheter in patients ventilated with a support mode and breathing spontaneously. Two, often used balloon catheters will be tested.

SECONDARY OUTCOMES:
The difference of optimal filling volume in spontaneously breathing and in passive ventilation (in cmH2O) | 45 minutes
  After measurements of the esophageal balloon were done during spontaneously breathing patients, measurements were done during mandatory ventilation while patient is passive. The measurements are the values and the optimal filling volume of the esophageal balloon in spontaneously breathing and in a passive mode.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Schoe, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request with researchers.

REFERENCES:
- [Background] Mojoli F, Iotti GA, Torriglia F, Pozzi M, Volta CA, Bianzina S, Braschi A, Brochard L. In vivo calibration of esophageal pressure in the mechanically ventilated patient makes measurements reliable. Crit Care. 2016 Apr 11;20:98. doi: 10.1186/s13054-016-1278-5. PMID 27063290
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Yoshida T, Grieco DL, Brochard L, Fujino Y. Patient self-inflicted lung injury and positive end-expiratory pressure for safe spontaneous breathing. Curr Opin Crit Care. 2020 Feb;26(1):59-65. doi: 10.1097/MCC.0000000000000691. PMID 31815775